CLINICAL TRIAL: NCT04974515
Title: Adherence to Electrical Glossal In Situ Stimulation for Sleep Apnea
Brief Title: Adherence to Electrical Glossal In Situ Stimulation for Sleep Apnea (AEGIS Study)
Acronym: AEGIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Naresh Punjabi, Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20210068
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Low intensity application of eXciteOSA (Experimental): Participants will receive the eXciteOSA device intervention at low intensity application for 20 minutes per day for 6 consecutive weeks.
  Interventions: Device: eXciteOSA
- High intensity application of eXciteOSA (Active Comparator): Participants will receive the eXciteOSA device intervention at high intensity application for 20 minutes per day for 6 consecutive weeks.
  Interventions: Device: eXciteOSA

INTERVENTIONS:
Device: eXciteOSA — eXciteOSA is a device for improving genioglossus endurance through electrical stimulation

SUMMARY:
The purpose of this research is to assess how well people with mild obstructive sleep apnea (OSA) adhere to the eXciteOSA device and specifically examine whether adherence of the device is different with low versus high electrical stimulation. In addition, this research study will assess how well the device affects mild sleep apnea and if it improves sleepiness and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Ability to consent
3. Home sleep apnea test demonstrating mild obstructive sleep apnea.
4. Smartphone or tablet

Exclusion Criteria:

1. Current pacemaker, defibrillator, or neuro-stimulation device
2. No prior oropharyngeal surgery for sleep apnea
3. No implants, metal prostheses, dental braces, or soft tissue/bony ulcerations in the oral cavity
4. No prior use of mandibular advancement device (MAD) or continuous positive airway pressure (CPAP)
5. Heart failure (New York Heart Association Class 3 or 4; or ejection fraction < 45%)
6. Active coronary disease defined as an intervention (e.g., angioplasty, coronary artery bypass surgery) in the prior 6 months
7. Uncontrolled hypertension (BP > 160/100)
8. Clinician diagnosis of any chronic lung disease except asthma
9. Chronic fatigue syndrome or fibromyalgia
10. Self-reported current illicit drug use in the past 30 days
11. Self-reported use of marijuana or opiates in the past 30 days
12. Use of supplemental oxygen
13. Self-reported use of prescribed or over the counter sleeping medications in the past 30 days
14. Current pregnancy or intention of becoming pregnant
15. Oropharyngeal abnormalities (class 2 or class 3 malocclusion)
16. Periodic breathing (Cheyne Stoke respiration)
17. Central sleep apnea (central apnea index (CAI) > 5/h)
18. Investigator discretion
19. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Punjabi, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with mild sleep apnea recruited from sleep clinic and general community
Period: Overall Study
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.6) | 50.5 (14.8) | 52.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 17 | 19 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 28.9 (4.5) | 28.4 (5.2) | 28.6 (4.8)
Respiratory event index [Mean (Standard Deviation); unit: events/hr] | 12.0 (3.8) | 12.6 (3.7) | 12.3 (3.)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] | 10.3 (5.3) | 8.2 (5.8) | 9.3 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Days Device Was Used
Description: Adherence level will be reported as the mean number of days the eXciteOSA device was used.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Number analyzed (Participants) | 19 | 21
Days | 38.0 (8.3) | 38.4 (7.4)

2. Secondary Outcome: Mean Respiratory Event Index (REI)
Description: The mean respiratory event index (events/hr) will be evaluated using a home sleep apnea test. A higher respiratory event index (REI) indicates greater frequency of abnormal breathing during sleep.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: events/hr
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Number analyzed (Participants) | 19 | 21
events/hr | 12.6 (1.2) | 9.6 (1.2)

3. Secondary Outcome: Epworth Sleepiness Scale (ESS) Scores
Description: Self-reported ESS questionnaire has a total score ranging from 0-24 with the higher score indicating greater daytime sleepiness.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Number analyzed (Participants) | 19 | 21
score on a scale | 9.4 (5.4) | 6.9 (4.3)

4. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Self-reported PSQI has a total score ranging from (0) to (21) with the higher score indicating worse sleep quality.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Number analyzed (Participants) | 19 | 21
score on a scale | 7.2 (4.3) | 5.5 (2.7)

5. Secondary Outcome: Short Form-20 (SF-20) Scores
Description: Self reported SF-20 has a total score ranging from 0-100 with the higher score indicating better quality of life.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Number analyzed (Participants) | 19 | 21
score on a scale | 76.6 (28.5) | 86.5 (15.0)

6. Secondary Outcome: Quality of Life as Measured by EuroQol Score
Description: Self-reported quality of life based on the EuroQoL has a total score ranging from 0 to 100 with the higher score indicating better quality of life
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Number analyzed (Participants) | 19 | 21
score on a scale | 0.88 (0.13) | 0.84 (0.08)

7. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Questionnaire Scores
Description: Self-reported WPAI questionnaire has a total score ranging from 0-20 the higher score indicating greater impairment daily activities.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Number analyzed (Participants) | 19 | 21
score on a scale | 1.0 (4.2) | 9.5 (17.2)

8. Secondary Outcome: Snoring Visual Analog Scores
Description: Partner reported Snoring visual analog has a total score ranging from 0-100 with the higher score indicating greater degree of snoring.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Number analyzed (Participants) | 19 | 21
score on a scale | 50.3 (22.0) | 42.5 (27.4)

9. Secondary Outcome: Number of Participants Accepting Long Term Treatment
Description: Number of participants reporting acceptance of long term treatment will be reported
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
Number analyzed (Participants) | 19 | 21
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Low Intensity Application of eXciteOSA | High Intensity Application of eXciteOSA
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04974515/Prot_SAP_000.pdf